CLINICAL TRIAL: NCT05332223
Title: The Epidemiological Characteristics of Sleep Disordered Breathing in Patients With Reduced or Preserved Ejection Fraction Congestive Heart Failure
Brief Title: The Epidemiology of Sleep Disordered Breathing in Patients With Congestive Heart Failure
Status: Completed | Type: Observational
Sponsor: Ministry of Health, Malaysia (Other Government)
Responsible Party: Principal Investigator, ALBERT ANTHONY, Pulmonologist, Ministry of Health, Malaysia
Other Study IDs: NMRR ID-22-00210-Y9W (IIR)
Record Dates: First submitted 2022-04-04; First posted 2022-04-18 (Actual); Last update posted 2024-02-15 (Actual); Status verified 2024-02

CONDITIONS: Chronic Heart Failure; Sleep Disorder
Keywords: Chronic Heart Failure; Sleep Disorder
MeSH Terms: conditions — Sleep Wake Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Chronic Heart Failure Patients: All patients in our specialised heart failure clinic will be screened by the investigator/s.
  Interventions: Diagnostic Test: Full Polysomnography

INTERVENTIONS:
Diagnostic Test: Full Polysomnography — Overnight PSG will be conducted using Alice version 6 system (Respironics, Pittsburgh, PA, USA). During PSG, the following variables will be monitored and captured. Sleep staging using electroencephalogram (four channels: C3-A2, C4-A1, O1-A2, O2-A1), electrooculogram (two channels: LOC-A2, ROC-A1), electromyogram (two channels: submental and anterior tibialis muscles). Respiratory effort using inductive plethysmograph sensors to detect thoracoabdominal movements. Oro-nasal airflow using pressure flow transducer and thermistor. Oxygen saturation using pulse oximetry and cardiac rhythm using electrocardiography. Other parameters that will also be monitored includes body position, presence of snoring and end tidal CO2 (EtCO2) measurement to detect hypercapnia. The attended PSG will be conducted in the sleep laboratory in Respiratory Unit, Hospital Taiping

SUMMARY:
This research will be one of the first hospital-based studies to comprehensively evaluate the epidemiological characteristics of sleep disordered breathing (SDB) in patients with Congestive Heart Failure (CHF). This prospective, observational cohort, single center study will include all consecutive CHF outpatients from the specialized heart failure clinic in Medical Department, Hospital Taiping, Malaysia irrespective of preserved or depressed Left Ventricular Ejection Fraction (LVEF). All participants will be subjected to an attended in-laboratory polysomnogram (PSG). It is anticipated the frequency and types of SDB to be variable compared to western data as this subject remains understudied in the South East Asian population. This research utilizes PSG rather than Portable Sleep Testing (PST) as seen in preceding studies for the diagnosis of SDB to prevent underdiagnosing SDBs and clearly distinguishing Obstructive Sleep Apnea (OSA) and Central Sleep Apnea (CSA).

DETAILED DESCRIPTION:
The epidemiology of SDB in CHF has not been studied in a South East Asian population. The results from studies conducted in USA and Europe on the prevalence of SDB in CHF may not be applicable to these patients for various reasons. Firstly, a diverse and multi -ethnic population in South East Asia may have an impact on the occurrence of SDB due to varying craniofacial morphological appearances, differences in levels of obesity and respiratory chemosensitivity. Additionally, the disparity in health services and the socio-economic differences between developed countries in the west and developing nations in South East Asia may have an impact on pharmacotherapy of CHF affecting the frequency and severity of SDB in these patients.

This research studies the epidemiological characteristics of SDB in non-selected, consecutive and consenting patients with CHF in the heart failure clinic as studying highly selected patients with clinical characteristics and risk factors of SBD may overestimate the prevalence. As patients with SDB in CHF may lack subjective EDS and assessment tools are unreliable in predicting SDB in CHF patients, the investigators wish to identify clinical predictors in this cohort of patients. It is anticipated there may be differences in this aspect when compared to patients in the western population and the investigators hope to obtain some understanding on the gender differences for SDB that has been reported in prior studies as well. The utility of attended in laboratory PSG as a diagnostic tool for all consecutive patients with CHF will prevent underestimation of AHI and clearly distinguish OSA and CSA based on standard definitions.

The prevalence of SDB in preserved ejection fraction CHF is understudied globally and the investigators wish to include preserved ejection fraction CHF patients apart from depressed ejection fraction CHF patients in this study. SDB presents as a treatment opportunity for patients with CHF but first the disorder has to be suspected and diagnosed. Initiation of nocturnal ventilation following diagnosis may treat the SDB and improve the prognosis of CHF.

ELIGIBILITY:
Inclusion Criteria:

* All patients with CHF regardless of LVEF Participants need to be older than 18 years old and is able to understand study information and give informed consent

Exclusion Criteria:

* Patients who had been diagnosed with SDB or is treated with any form of Positive Airway Pressure (PAP) therapy prior to this will be excluded from this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All consecutive adult patients under follow-up in Heart Failure Clinic, Hospital Taiping during the period 1 April 2022 - 31 December 2024
Sampling Method: Non-Probability Sample
Enrollment: 116 (Actual)
Dates: Start 2022-04-15 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2023-12-31 (Actual)

PRIMARY OUTCOMES:
Presence of Sleep Disordered Breathing | through study completion, an average of 2 years
  Present or Absent
Type of Sleep Disordered Breathing | through study completion, an average of 2 years
  Obstructive or Central Sleep Apnoea

CONTACTS AND LOCATIONS:
Overall Officials: ALBERT IRUTHIARAJ L. ANTHONY, MBBS, Principal Investigator — HOSPITAL TAIPING
Locations (1):
- Hospital Taiping, Taiping, Perak, Malaysia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Arzt M, Young T, Finn L, Skatrud JB, Ryan CM, Newton GE, Mak S, Parker JD, Floras JS, Bradley TD. Sleepiness and sleep in patients with both systolic heart failure and obstructive sleep apnea. Arch Intern Med. 2006 Sep 18;166(16):1716-22. doi: 10.1001/archinte.166.16.1716. PMID 16983049
- [Background] Arzt M, Woehrle H, Oldenburg O, Graml A, Suling A, Erdmann E, Teschler H, Wegscheider K; SchlaHF Investigators. Prevalence and Predictors of Sleep-Disordered Breathing in Patients With Stable Chronic Heart Failure: The SchlaHF Registry. JACC Heart Fail. 2016 Feb;4(2):116-125. doi: 10.1016/j.jchf.2015.09.014. Epub 2015 Dec 9. PMID 26682790
- [Background] Collop NA, Anderson WM, Boehlecke B, Claman D, Goldberg R, Gottlieb DJ, Hudgel D, Sateia M, Schwab R; Portable Monitoring Task Force of the American Academy of Sleep Medicine. Clinical guidelines for the use of unattended portable monitors in the diagnosis of obstructive sleep apnea in adult patients. Portable Monitoring Task Force of the American Academy of Sleep Medicine. J Clin Sleep Med. 2007 Dec 15;3(7):737-47. PMID 18198809
- [Background] Chan J, Sanderson J, Chan W, Lai C, Choy D, Ho A, Leung R. Prevalence of sleep-disordered breathing in diastolic heart failure. Chest. 1997 Jun;111(6):1488-93. doi: 10.1378/chest.111.6.1488. PMID 9187161
- [Result] Joynt KE, Jha AK. Who has higher readmission rates for heart failure, and why? Implications for efforts to improve care using financial incentives. Circ Cardiovasc Qual Outcomes. 2011 Jan 1;4(1):53-9. doi: 10.1161/CIRCOUTCOMES.110.950964. Epub 2010 Dec 14. PMID 21156879
- [Derived] Lourdesamy Anthony AI, Abdul Rani R. The epidemiological characteristics of sleep disordered breathing in congestive heart failure: A prospective, single centre study in Southeast Asia. J R Coll Physicians Edinb. 2024 Mar;54(1):18-25. doi: 10.1177/14782715241239704. Epub 2024 Mar 20. PMID 38509698